CLINICAL TRIAL: NCT05615792
Title: Observational Cohort of The Effects of Clinical Indicators, Drug Use and Genotypes on The Clinical Prognosis of COVID-19 Patients in Hubei Province
Brief Title: Observational Cohort of COVID-19 Patients in Hubei Province
Acronym: OCCP-HP
Status: Completed | Type: Observational
Sponsor: Dao Wen Wang (Other)
Responsible Party: Sponsor-Investigator, Dao Wen Wang, Prof., Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-COVID
Record Dates: First submitted 2022-11-10; First posted 2022-11-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: 2019 Novel Coronavirus Disease
Keywords: COVID-19; SARS-CoV-2; Risk Factors; Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with coronavirus disease 2019 (COVID-19): Patients diagnosed with COVID-19 in Hubei Province
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study intends to use the relevant case data of COVID-19 in Hubei Province, using big data processing and mining methods to evaluate the effects of clinical indicators, drug use and genes on the clinical prognosis of COVID-19 patients, so as to provide a theoretical basis for the treatment of these diseases and reduce the mortality.

DETAILED DESCRIPTION:
Hubei Province, as the forefront of the fight against epidemic, has the largest number of patients infected with SARS-CoV-2 and the highest quality medical data. However, so far, these data have not been fully analyzed, if these data can not be mined and used, it will be a great loss to the whole human race. By fully mining and analyzing these data, we can sum up a large number of experiences related to COVID-19, summarize various laws of this kind of disease, and provide clinical evidence based on large samples for the research of this disease, eventually contribute China's experience to the global fight against the epidemic.

Based on the above background, this study intends to use the relevant case data of COVID-19 in Hubei Province, using big data processing and mining methods to evaluate the effects of clinical indicators, drug use and genes on the clinical prognosis of COVID-19 patients, so as to provide a theoretical basis for the treatment of these diseases and reduce the mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, regardless of gender;
2. A history of epidemiology, including travel or residence in high-risk areas or other communities with case reports within 14 days before the onset of the disease, or have a history of contact with novel coronavirus infection (those who are positive for nucleic acid tests); or patients with fever or respiratory symptoms from the community with case reports; or aggregative onset;
3. Corresponding clinical manifestations, including respiratory symptoms such as fever, with typical imaging features of COVID-19, normal or decreased white blood cell count and decreased lymphocyte count in the early stage of the disease;
4. Clear etiological evidence, including real-time fluorescent RT-PCR detection of novel coronavirus nucleic acid positive, or viral gene sequencing, is highly homologous to novel coronavirus.

Exclusion Criteria:

Patients who meet any of the following criteria cannot be enrolled in this study:

1. Patients refused to participate in this study;
2. According to the researchers, patients are unable to complete this study or comply with the requirements of this study (due to management or other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a hospital-based observational study initiated by Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology. Trained researchers are responsible for screening and joining the group. About 6,8000 COVID-19 patients in Hubei Province were expected to be included in this study. Patients enrolled in the group will undergo baseline survey and follow-up according to the program.
Sampling Method: Probability Sample
Enrollment: 68000 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 2 years
  Numbers and dates of death in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li D, He W, Yu B, Wang DW, Ni L. NT-proBNP ratio is a potential predictor for COVID-19 outcomes in adult Chinese patients: a retrospective study. Sci Rep. 2024 Mar 11;14(1):5906. doi: 10.1038/s41598-024-56329-2. PMID 38467760
- [Derived] Xu K, He W, Yu B, Zhong K, Zhou D, Wang DW. Beneficial Effects of Angiotensin II Receptor Blockers on Mortality in Patients with COVID-19: A Retrospective Study from 2019 to 2020 in China. Cardiovasc Drugs Ther. 2025 Feb;39(1):63-74. doi: 10.1007/s10557-023-07494-5. Epub 2023 Aug 11. PMID 37566218